CLINICAL TRIAL: NCT03038763
Title: Vertical Transmission of Hepatitis C in Adult Children of Female Baby Boomers
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 826229
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C; Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers: Black or white mothers who have or have had hepatitis C and were born between 1945-1964. Participants must have at least one child over the age of 18.
  Interventions: Other: Eligibility Screening
- Adult Children: Adult children of Black or white mothers who have or have had hepatitis C and were born between 1945-1964. From speaking with these mothers, it must be possible that participants were exposed to hepatitis C virus while in the womb.
  Interventions: Diagnostic Test: HCV test

INTERVENTIONS:
Other: Eligibility Screening — Investigators will call eligible mothers to screen for the possibility that eligible mothers may have passed HCV on to adult children. Investigators will consent these mothers to contact the adult child(ren), as the child(ren) must be informed of the mother's HCV status, if not already known.
  Groups: Mothers
Diagnostic Test: HCV test — Adult children will be invited to Penn or a Penn affiliate to have labwork, testing HCV antibody and HCV quant. If the quant comes back positive, investigators will also test genotype and fibrosure.
  Groups: Adult Children

SUMMARY:
The investigators aim to determine the prevalence of hepatitis C in the adult children of female baby boomers. During the years baby boomers were becoming pregnant, hepatitis C testing was either not available or was not standard of care. Because of this, participants' children may be unaware of participants' risk of hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

Mothers:

* Born between 1/1/45-12/31/64
* Black or white race
* Active or prior infection with hepatitis C
* Have at least one living adult child over the age of 18

Children:

* ≥18 years of age
* Born to mother with current or prior HCV infection, with likely timing of HCV acquisition prior to or during pregnancy
* Mother gave informed consent for child to be approached for study participation

Exclusion Criteria:

Mothers:

- Unwilling to disclose hepatitis C status to children

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult children of women born between 1945-1965 who have or have had hepatitis C Women born between 1945-1965 who have or have had hepatitis C
  Investigators will only be recruiting subjects who are black or white as hepatitis C is most common in these two populations. Using these populations maximizes the generalizability of our results. HCV is not only significantly less common among Asian women and women of other races, but these women also represent a minority of the patient population at Penn.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
HCV prevalence | Within 1 week of labwork at first study visit
  Prevalence of HCV in adult children of female baby boomers who have or have had HCV

SECONDARY OUTCOMES:
Liver fibrosis | Within 2 weeks of diagnosis of HCV
  Level of liver fibrosis (detected through fibrosure test) found in adult children diagnosed as HCV-positive
HCV genotype | Within 6 weeks of diagnosis of HCV
  HCV genotype for adult children diagnosed as HCV-positive

CONTACTS AND LOCATIONS:
Overall Officials: David Goldberg, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rein DB, Smith BD, Wittenborn JS, Lesesne SB, Wagner LD, Roblin DW, Patel N, Ward JW, Weinbaum CM. The cost-effectiveness of birth-cohort screening for hepatitis C antibody in U.S. primary care settings. Ann Intern Med. 2012 Feb 21;156(4):263-70. doi: 10.7326/0003-4819-156-4-201202210-00378. Epub 2011 Nov 4. PMID 22056542
- [Background] Voelker R. Birth cohort screening may help find hepatitis C cases. JAMA. 2012 Mar 28;307(12):1242. doi: 10.1001/jama.2012.337. No abstract available. PMID 22453559
- [Background] AASLD/IDSA HCV Guidance Panel. Hepatitis C guidance: AASLD-IDSA recommendations for testing, managing, and treating adults infected with hepatitis C virus. Hepatology. 2015 Sep;62(3):932-54. doi: 10.1002/hep.27950. Epub 2015 Aug 4. No abstract available. PMID 26111063
- [Background] Benova L, Mohamoud YA, Calvert C, Abu-Raddad LJ. Vertical transmission of hepatitis C virus: systematic review and meta-analysis. Clin Infect Dis. 2014 Sep 15;59(6):765-73. doi: 10.1093/cid/ciu447. Epub 2014 Jun 13. PMID 24928290
- [Background] Kuncio DE, Newbern EC, Johnson CC, Viner KM. Failure to Test and Identify Perinatally Infected Children Born to Hepatitis C Virus-Infected Women. Clin Infect Dis. 2016 Apr 15;62(8):980-5. doi: 10.1093/cid/ciw026. Epub 2016 Jan 20. PMID 26797211
- [Background] Kabiri M, Jazwinski AB, Roberts MS, Schaefer AJ, Chhatwal J. The changing burden of hepatitis C virus infection in the United States: model-based predictions. Ann Intern Med. 2014 Aug 5;161(3):170-80. doi: 10.7326/M14-0095. PMID 25089861
- [Background] Mast EE, Hwang LY, Seto DS, Nolte FS, Nainan OV, Wurtzel H, Alter MJ. Risk factors for perinatal transmission of hepatitis C virus (HCV) and the natural history of HCV infection acquired in infancy. J Infect Dis. 2005 Dec 1;192(11):1880-9. doi: 10.1086/497701. Epub 2005 Oct 28. PMID 16267758
- [Background] Poynard T, Imbert-Bismut F, Munteanu M, Messous D, Myers RP, Thabut D, Ratziu V, Mercadier A, Benhamou Y, Hainque B. Overview of the diagnostic value of biochemical markers of liver fibrosis (FibroTest, HCV FibroSure) and necrosis (ActiTest) in patients with chronic hepatitis C. Comp Hepatol. 2004 Sep 23;3(1):8. doi: 10.1186/1476-5926-3-8. PMID 15387887
- [Background] Poynard T, Imbert-Bismut F, Munteanu M, Ratziu V. FibroTest-FibroSURE: towards a universal biomarker of liver fibrosis? Expert Rev Mol Diagn. 2005 Jan;5(1):15-21. doi: 10.1586/14737159.5.1.15. PMID 15723588
- [Background] Patel K, Benhamou Y, Yoshida EM, Kaita KD, Zeuzem S, Torbenson M, Pulkstenis E, Subramanian GM, McHutchison JG. An independent and prospective comparison of two commercial fibrosis marker panels (HCV FibroSURE and FIBROSpect II) during albinterferon alfa-2b combination therapy for chronic hepatitis C. J Viral Hepat. 2009 Mar;16(3):178-86. doi: 10.1111/j.1365-2893.2008.01062.x. Epub 2008 Oct 24. PMID 19175870
- [Background] Sebastiani G, Castera L, Halfon P, Pol S, Mangia A, Di Marco V, Pirisi M, Voiculescu M, Bourliere M, Alberti A. The impact of liver disease aetiology and the stages of hepatic fibrosis on the performance of non-invasive fibrosis biomarkers: an international study of 2411 cases. Aliment Pharmacol Ther. 2011 Nov;34(10):1202-16. doi: 10.1111/j.1365-2036.2011.04861.x. Epub 2011 Oct 9. PMID 21981787
- [Background] Poynard T, Bedossa P, Opolon P. Natural history of liver fibrosis progression in patients with chronic hepatitis C. The OBSVIRC, METAVIR, CLINIVIR, and DOSVIRC groups. Lancet. 1997 Mar 22;349(9055):825-32. doi: 10.1016/s0140-6736(96)07642-8. PMID 9121257
- [Background] Thein HH, Yi Q, Dore GJ, Krahn MD. Estimation of stage-specific fibrosis progression rates in chronic hepatitis C virus infection: a meta-analysis and meta-regression. Hepatology. 2008 Aug;48(2):418-31. doi: 10.1002/hep.22375. PMID 18563841